CLINICAL TRIAL: NCT07158489
Title: Protocol SAKK 18/ 25 Overcoming Resistance to Immunotherapy Combining Gemcitabine With Ivonescimab in Advanced NSCLC Progressing on Immune Checkpoint Inhibitors: A Multicenter, Single-arm, Open-label Phase II Trial (ORIGIN2)
Brief Title: Overcoming Resistance to Immunotherapy Combining Gemcitabine With Ivonescimab in Advanced NSCLC
Acronym: ORIGIN2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 18/25
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: NSCLC; NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: advanced NSCLC; immune checkpoint inhibitors; Resistance to immunotherapy; Gemcitabine and Ivonescimab; Gemcitabine; Ivonescimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine + Ivonescimab in Advanced NSCLC Resistant to Immunotherapy (Experimental)
  Interventions: Drug: Gemcitabine + Ivonescimab

INTERVENTIONS:
Drug: Gemcitabine + Ivonescimab — The trial combines two Investigational Medicinal Products (IMPs):
  * Gemcitabine, either alone or in combination regimens, is the standard of care (SoC) for several solid tumors, such as advanced or metastatic non-small cell lung cancer (mNSCLC).
  * Ivonescimab is developed for cancer immunotherapy. Ivonescimab binds to human vascular endothelial growth factor (VEGF) which is involved in tumor angiogenesis, and to human programmed cell death 1 (PD-1) that is a cell surface receptor expressed primarily on activated T cells and acts to inhibit their activation.

SUMMARY:
This Phase II clinical trial (investigates the efficacy of combining gemcitabine, a chemotherapy agent, with ivonescimab, a bispecific PD-1/VEGF antibody, in patients with advanced non-small cell lung cancer (NSCLC) who have experienced disease progression following chemoimmunotherapy (CIT). Lung cancer remains the leading cause of cancer-related death globally, and treatment options after CIT failure are limited. Gemcitabine has demonstrated immunostimulatory properties, including enhanced T-cell infiltration and reduced immunosuppressive cell populations, which may synergize with immune checkpoint inhibitors. Ivonescimab targets both PD-1 and VEGF pathways, potentially enhancing antitumor immune responses and inhibiting tumor angiogenesis. The trial aims to evaluate the objective response rate (ORR) according to RECIST v1.1 criteria. The combination therapy is expected to offer a novel and effective treatment strategy for patients with relapsed NSCLC, addressing a significant unmet medical need.

DETAILED DESCRIPTION:
Lung cancer is the most frequently diagnosed cancer worldwide, with approximately 2.5 million new cases and 1.8 million deaths annually. Most cases are diagnosed at an advanced stage, necessitating systemic therapy. Although chemoimmunotherapy (CIT) has improved outcomes, disease progression remains inevitable, and second-line treatments offer limited efficacy. Gemcitabine, a cytidine analogue, interferes with DNA synthesis and exhibits immunomodulatory effects, including increased effector T-cell infiltration and reduced regulatory T-cell activity. Preclinical studies have shown that gemcitabine enhances antitumor immune responses when combined with immune checkpoint inhibitors (ICIs), such as anti-PD-1 antibodies.

Ivonescimab (AK112/SMT112) is a bispecific antibody targeting PD-1 and VEGF, designed to simultaneously modulate immune and angiogenic pathways. It binds to PD-1 on activated T cells and VEGF involved in tumor angiogenesis. The combination of gemcitabine and ivonescimab is hypothesized to synergistically improve antitumor activity in patients with advanced NSCLC who have progressed after CIT.

Preclinical evidence from mouse models of mesothelioma demonstrated that combining gemcitabine with immunotherapy significantly increased survival and lymphocyte infiltration at the tumor site. This effect was negated by dexamethasone, highlighting the importance of immune modulation. Clinical observations in mesothelioma patients further support the potential of this combination.

Gemcitabine is a standard of care (SoC) for several solid tumors, including NSCLC. Its immunostimulatory properties make it a suitable candidate for combination with ICIs. Ivonescimab has shown superior efficacy compared to pembrolizumab in PD-L1+ NSCLC patients in first-line settings. Despite ongoing trials exploring similar combinations, none have investigated gemcitabine with ivonescimab.

This Phase II trial aims to assess the antitumor activity of gemcitabine combined with ivonescimab in patients with advanced NSCLC who have limited therapeutic options. Gemcitabine will be administered according to standard treatment recommendations, while ivonescimab will be given at 20 mg/kg every three weeks (q3w), consistent with previous trials.

The primary objective is to evaluate the objective response rate (ORR) based on RECIST v1.1 criteria, with independent response review. The study is inclusive across sex, gender, and ethnicity, and all materials will use gender-inclusive language. A positive outcome may support the adoption of this combination as a new standard treatment for relapsed NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling all of the following inclusion criteria are eligible for the trial:
* Written informed consent according to Swiss law and ICH GCP E6 regulations before registration and prior to any trial specific procedures including patient screening.
* Confirmed squamous or non-squamous mNSCLC stage IIIB-IV (based on 9th edition Tumor-Node-Metastasis (TNM) classification of lung cancers with disease recurrence or progression during or after one or more prior immunotherapy or CIT regimens for metastatic disease.
* Patients with treated and stable central nervous system (CNS) metastases are eligible, if:

  * Previous CNS-directed therapy has been completed at least 4 weeks prior to treatment start.
  * No evidence of progression after completion of CNS-directed therapy as ascertained by clinical examination and brain imaging with Magnetic Resonance Imaging (MRI) or CT.25
* Patients with known HIV-infection are eligible, if:

  * CD4+ T-cell counts are ≥ 350 cells/µl
  * No history of AIDS-defining opportunistic infection within past 12 months
  * Patient agrees to concomitant antiretroviral therapy (ART) if not currently on ART, or is on ART for ˃ 4 weeks and has a HIV viral load ˂ 400 copies/ml.26
* Patients with a previously treated malignancy are eligible if this is clinically stable and does not require concurrent tumor-directed treatment.

Exception: patients suffering from prostate cancer under hormonal ablation therapy (hormone sensitive disease).

* Patients with measurable disease according to RECIST v1.1.
* Availability of newly collected or archival (maximum 3 months) samples for TR prior to treatment initiation.
* Age ≥ 18 years
* ECOG performance status 0-2.
* Adequate bone marrow function: absolute neutrophil count ≥ 1.5 x 109/l, platelet count ≥ 100 x 109/l, hemoglobin ≥ 90 g/l.

6.1.11 Adequate hepatic function: total bilirubin ≤ 1.5 x upper limit of normal ([ULN]; except for patients with Gilbert's disease ≤ 3.0 x ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN, or ≤ 5 x ULN for patients with hepatic metastasis.

* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 40 ml/min/1.73 m2 (according to the Chronic Kidney Disease Epidemiology Collaboration) abbreviated formula CKD-EPI formula.
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must use highly effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 6 months after the last dose of investigational drug . A negative serum or urine pregnancy test before starting trial treatment is required for all women of childbearing potential.
* Men agree not to donate sperm or father a child during trial treatment and until 6 months after the last administration of investigational drug.
* Patients give their consent to participate in TR projects and providing the mandatory samples.

Exclusion Criteria:

* Symptomatic brain metastases.
* Prior treatment with gemcitabine in combination with immunotherapies.
* Tumor progression within the first 8 weeks from start of first-line treatment.
* Activating EGFR or ALK mutations.
* Concomitant use of other anti-cancer drugs or radiotherapy.
* Major surgery within 1 month prior to treatment start.
* Known history of any uncontrolled active systemic infection requiring intravenous antimicrobial treatment.
* Known history of tuberculosis, primary immunodeficiency, allogeneic tissue/solid organ transplant, or receipt of live attenuated vaccine.
* History of interstitial lung disease or severe pneumonitis.
* Concomitant use of corticosteroids as premedication for gemcitabine therapy.
* Concomitant or prior use of immunosuppressive medication such as interferon or methotrexate within 28 days prior to trial treatment start, with the exceptions of local (i.e., intranasal, inhaled and topical) corticosteroids.
* Major blood vessel tumor invasion.
* Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to study treatment initiation.
* Unstable angina, myocardial infarction, congestive heart failure (NYHA classification Grade ≥2;27) or vascular disease (e.g., aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to study treatment initiation, or other cardiac impairment that may affect the safety evaluation of the study drug (e.g., poorly controlled arrhythmias, myocardial ischemia).
* History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to study treatment initiation.
* History of arterial thromboembolic event, venous thromboembolic event of Grade ≥3 as specified in NCI CTCAE v5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to study treatment initiation.
* Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks prior to study treatment initiation.
* History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to study treatment initiation.
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information or to the Investigator's Brochure (IB).
* Known or suspected hypersensitivity to gemcitabine or ivonescimab or to any component of the trial drugs.
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to registration, including but not limited to:

  * Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots).

Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.

* Nasal bleeding /epistaxis (bloody nasal discharge is allowed).
* Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to registration is not allowed. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time is within therapeutic limits according to the medical standard of the enrolling institution.

  * Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic pressure ≥ 100 mmHg after oral antihypertensive therapy.
  * Active autoimmune or lung disease requiring systemic therapy (e.g., with disease modifying drugs, prednisone >10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to registration, however the following will be allowed:
* Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
* Intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections is permitted.

  * Has pre-existing peripheral neuropathy that is ≥ Grade 2 by NCI CTCAE v5.0.
  * Uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic.

Note: Patients managed with indwelling catheters (e.g., PleurX) are allowed.

* History of non-infectious pneumonia requiring systemic corticosteroids, or current interstitial lung disease.
* Active or prior history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea).
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST v1.1 | At the end of trial treatment, up to 2 years from registration.
  ORR according to RECIST v1.1 is defined as the proportion of patients, whose best overall response is either complete response (CR) or partial response (PR) achieved before disease progression according to RECIST v1.1 or start of a subsequent anti-cancer treatment whichever occurs first.
  Patients with CR or PR as best observed response will be considered as success; otherwise as failures for this endpoint.
  Patients without any tumor assessment or with non-evaluable response (NE) during trial treatment will be considered as failures for this endpoint.
  The primary analysis will be based on the results from the Independent Response Review.

SECONDARY OUTCOMES:
Duration of response (DoR) according to RECIST v1.1 | From first response up to 2 years from treatment start.
  DoR according to RECIST v1.1 is defined as the time from the first documentation of CR or PR (whichever occurs first) until disease progression according to RECIST v1.1 or death due to any cause. Patients not experiencing an event at the time of analysis and those starting a subsequent anticancer treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent anti-cancer treatment, if any.
  This endpoint will be calculated for the subgroup of patients achieving CR or PR.
  The analysis of this endpoint will be based on the independent response review.
Progression-free Survival (PFS) according to RECIST v1.1 | From first dose of ivonescimab/gemcitabine, up to 2 years from treatment start.
  PFS according to RECIST v1.1 is measured as the time from the first dose of ivonescimab/gemcitabine until disease progression according to RECIST v1.1 or death due to any cause.
  Patients not experiencing an event at the time of analysis and those receiving a subsequent anti-cancer treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent anti-cancer treatment, if any.
  The analysis of this endpoint will be based on the independent response review.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Curioni-Fontecedro, Prof, Study Chair — Cantonal Hospital Fribourg / University of Fribourg
Locations (7):
- Switzerland (7):
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - IOSI Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Hôpital Fribourgeois - Hôpital Cantonal, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No